CLINICAL TRIAL: NCT05971290
Title: Effects of Continuous Positive Airway Pressure on Peripheral Oxygen Saturation, Work of Breathing, and Exercise Tolerance at Altitude
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0468
Record Dates: First submitted 2023-07-06; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Hypoxemia; Altitude Hypoxia
MeSH Terms: conditions — Hypoxia; Altitude Sickness | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Positive Airway Pressure use (Experimental)
  Interventions: Device: Continuous positive airway pressure
- Ambient air (Sham Comparator)
  Interventions: Device: Ambient air

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure administered by face mask
  Arms: Continuous Positive Airway Pressure use
Device: Ambient air — Air (fraction of inspired oxygen) at 14000 feet in elevation
  Arms: Ambient air

SUMMARY:
Dyspnea and exercise intolerance are well known to travelers who have experienced time at high elevations, greater than 2500 meters (8200 feet). As individuals ascend to higher elevations, oxygen saturations significantly decrease as the partial pressure of oxygen decreases. Additionally, many individuals develop subclinical cases of high altitude pulmonary edema (HAPE), which may worsen hypoxemia and decrease exercise performance. While dyspnea and exercise intolerance are usually self-limiting and improve with rest, some individuals experience severe symptoms that prevent safe evacuation to lower elevation.

Individuals experiencing high altitude dyspnea, subclinical HAPE, or clinical HAPE will see improvements in symptoms and SpO2 when receiving supplemental oxygen, however this requires heavy and unwieldy tanks that make it difficult to carry across irregular terrain. Additionally, given the often-remote conditions where supplemental oxygen is needed, it is often difficult to replenish supplies. Other devices, such as the portable hyperbaric chamber (often referred to as Gamow bag), can temporarily improve dyspnea and oxygen saturation at high and extreme altitudes without the use of oxygen tanks. This device also carries some of the same disadvantages as supplemental oxygen, however, as the bag is also heavy and patients are not ambulatory while using the device.

Similar to supplemental oxygen and the portable hyperbaric chamber, there is some evidence that CPAP may improve SpO2 and dyspnea at high and extreme altitudes. CPAP has already demonstrated significant efficacy in reducing symptoms of acute mountain sickness (AMS) when used in the field. At the time these small studies were conducted, CPAP therapy carried similar disadvantages in weight and portability. In recent years, however, CPAP devices have become increasingly lightweight and portable, with recent models weighing less than 1 kilogram (2.2 pounds). These devices are often powered by batteries, which themselves are light and easy to carry, and can be charged in the field using either a generator or foldable solar panels. These newer features of CPAP devices overcome some of the previous disadvantages that have limited its potential uses. CPAP devices can easily be carried across difficult terrain directly to individuals suffering from altitude-related symptoms, to be used as a rescue device until definitive care is available. Its portability not only allows for easy delivery to a patient, but also may allow for a patient to experience enough symptom relief to walk themselves down to lower elevation, greatly improving speed and resource utilization involved in high altitude rescues.

In previous studies, CPAP devices have been found to be effective and safe to use in high and extreme altitude locations. While a few pilot studies have assessed CPAP's utility in treating dyspnea and SpO2 at altitude, these studies were done at rest. While one study showed improved symptoms and SpO2 in normobaric and hypobaric hypoxia, the study was limited by its lack of real-world condition, and its authors suggested further study in field and extreme environmental conditions. Additional investigation is needed to determine whether or not CPAP is an effective tool in the field to improve SpO2, dyspnea, and exercise tolerance in individuals traveling at high elevations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults (age 18-70)
* Living at lower elevation (<2500m or 8200ft)

Exclusion Criteria:

* Age > 70 or age < 18.
* History of chronic respiratory conditions (asthma, COPD, ILD)
* Obstructive sleep apnea (if currently using nighttime CPAP)
* Congestive heart failure, coronary artery disease
* History of myocardial infarction
* History of HAPE
* Neurologic disorder
* Cognitive disorder
* Altered mental status
* Pregnancy
* Current use of supplemental oxygen
* Impaired mobility
* Excessive facial hair
* Claustrophobia.
* Current use of altitude-related illness prophylaxis medications
* Current use of anticoagulant medications
* Current use of calcium channel blockers medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-22 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral oxygen saturation | 1 day
  SpO2 measurement in percentage
Respiratory rate | 1 day
  Breaths/minute
Heart rate | 1 day
  Heartbeats/minute

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Strickland, MD, Principal Investigator — UC Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT05971290/ICF_000.pdf